CLINICAL TRIAL: NCT01871883
Title: Distribution and Expression of Non-neuronal Transient Receptor Potential (TRPV) Ion Channels in Sensitive Skin Syndrome.
Brief Title: TRPV Expression in Subjects With Sensitive Skin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Dermatology Research Director, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TRPV1SenSk
Record Dates: First submitted 2013-05-27; First posted 2013-06-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Sensitive Skin
Keywords: Sensitive skin; Transient potential receptor vanilloid 1; TRPV1; Transepidermal water loss; Skin Phototype; Lactic acid test; Skin irritancy tests

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensitive Skin (Experimental): Subjects with sensitive skin, diagnosed by the lactic acid stinging test. Skin biopsy Oral mucosa specimen
  Interventions: Procedure: Skin biopsy; Procedure: Oral mucosa specimen
- Non-sensitive skin (Active Comparator): Subjects without sensitive skin, determined by a negative lactic acid stinging test Skin biopsy Oral mucosa specimen
  Interventions: Procedure: Skin biopsy; Procedure: Oral mucosa specimen

INTERVENTIONS:
Procedure: Skin biopsy — Two skin biopsies will be taken with a 3 mm punch in the retroauricular area. The procedure will be done by an investigator, under aseptic and antiseptic conditions and under local anesthesia with lidocaine and epinephrine. The incision will be sutured with 6-0 Nylon, and the stitches will be removed after 5 days. One biopsy will be processed for immunohistochemistry, the other for RNA extraction and analysis.
  Other Names: Skin biopsy by punch
Procedure: Oral mucosa specimen — The sample for keratinocytes from oral mucosa will be taken with a Foam knife, which is a non-invasive procedure. It does not need anesthesia, and it does not leave scars. The procedure consists in gently brush the oral mucosa with the knife five times, and the material that will be obtained will be fixed in a PBS solution for RNA analysis.
  Other Names: Oral mucosa keratinocytes; Oral mucosa swap

SUMMARY:
Sensitive skin syndrome is defined as the presence of burning, itching or any other unpleasant sensation on the skin, due to physical, chemical or psychological factors. It is frequently a self-diagnosed condition, and there are no accurate tests to recognize or quantify it because of the individual variations in perception and intensity of the related symptoms. The most accepted physiopathogenic theory is the presence of an altered barrier function of epidermis. Also, changes in the pH of the stratum corneum have been found to induce skin sensitivity through the activation of the transient potential receptor vanilloid (TRPV) neuronal receptors.

TRPV1 has been found in human keratinocytes, although its physiologic role in the skin is not yet established. Their presence in keratinocytes and cutaneous nervous fibers suggests a role in the sensitive function of the epidermis. Since this receptors can be activated by low pH (< 5.9), which is also important for the development of sensitive skin, we hypothesized that an increase in the expression of these receptors can be the responsible for the syndrome.

DETAILED DESCRIPTION:
Sensitive skin syndrome is defined as the presence of burning, itching or any other unpleasant sensation on the skin, due to physical, chemical or psychological factors. It is frequently a self-diagnosed condition, and there are no accurate tests to recognize or quantify it because of the individual variations in perception and intensity of the related symptoms.

Although the pathogenesis of sensitive skin syndrome is not completely understood, the most accepted theory is the presence of an altered barrier function. Irritation results from the abnormal penetration of substances to deeper layers of the skin, where they can induce vasodilation and stimulate c-type neuronal fibers. Also, changes in the pH of the stratum corneum have been found to induce skin sensitivity through the activation of the transient potential receptor vanilloid (TRPV) neuronal receptors.

TRPV1 was first discovered in 1997, when it was identified as the specific receptor for capsaicin in a subgroup of nociceptors. It is a non-selective thermo-sensitive cationic channel that can be found in nerves from the central and peripheral nervous system, fibroblasts, smooth muscle, mast cells, endothelial cells, gastrointestinal, respiratory and urinary epithelial cells. TRPV1 can be activated by excessive heat (>42ºC), acidic pH (< 5.9), and also by endogenous substances such as N- arachidonoyl dopamine, leucotriene B, phospholipase C, and many others.

In 2001, the functional expression of TRPV1 was identified in human keratinocytes. Their physiologic role in the skin has not been completely understood, but they have been related to differentiation, proliferation, inflammation and homeostasis of the epidermal barrier. Their presence in keratinocytes and cutaneous nervous fibers suggests a role in the sensitive function of the epidermis. It has been proved that the stimulation of TRPV1 in neuronal cells can induce pruritus and burning sensation. In vitro studies have demonstrated that the exogenous stimulation of TRPV1 in keratinocytes induces the release of nitric oxide, ATP, dopamine, prostaglandins, and other pro-inflammatory substances that can act as paracrine mediators between keratinocytes and cutaneous nerve fibers. Therefore, there are scientific bases to hypothesize that an increase in the expression of these receptors can be the responsible for the sensitive skin syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Known response to the lactic acid stinging test
* Informed signed consent

Exclusion Criteria:

* Any dermatoses in the test area
* Use of topical medications in the test area
* Personal history of keloid or hypertrophic scarring
* Known allergy to lidocaine
* Know heart disease
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Expression of TRPV1 | Up to 1 year
  Determine the expression of TRPV1 in patients with sensitive skin

SECONDARY OUTCOMES:
TRPV1 and Sensitive Skin | Up to 1 year
  Correlate the expression of TRVP1 with the presence of sensitive skin syndrome
TRPV1 and skin phototype | Up to 1 year
  Identify variations in the expression of TRPV1 according to skin phototype
TRPV1 and barrier function | Up to 1 year
  Correlate the expression of TRPV1 with the transepidermal water loss as an indirect measure of barrier function.

OTHER OUTCOMES:
TRPV1 mRNA in biopsies | Up to 1 year
  Quantify the expression of mRNA of TRPV1 in epidermal keratinocytes obtained by skin biopsies through RT-PCR
TRPV1 in biopsies by immunohistochemistry | Up to 1 year
  Quantify the expression of TRPV1 in epidermal keratinocytes obtained by skin biopsies through immunohistochemistry
mRNA1 of TRPV1 in oral keratinocytes | Up to 1 year
  Quantify the expression of mRNA of TRPV1 in epidermal keratinocytes obtained from oral mucosa through RT-PCR
TRPV1 in oral keratinocytes by immunohistochemistry | Up to 1 year
  Quantify the expression of TRPV1 in epidermal keratinocytes obtained from oral mucosa through immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Ehnis-Pérez, MD, Principal Investigator — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"; Juan P Castanedo-Cázares, MD, Study Director — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"; Bertha Torres-Álvarez, MD, Study Chair — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Hernández-Blanco D, Castanedo-Cázares JP, Ehnis-Pérez A, Jasso-Ávila I, Conde-Salazar L, Torres-Álvarez B. Prevalence of sensitive skin and its biophysical response in a Mexican population. World J Dermatol 2013;2:1-7. doi:10.5314/wjd.v2.i1.1.
- [Background] Escalas-Taberner J, Gonzalez-Guerra E, Guerra-Tapia A. [Sensitive skin: a complex syndrome]. Actas Dermosifiliogr. 2011 Oct;102(8):563-71. doi: 10.1016/j.ad.2011.04.011. Epub 2011 Jul 14. Spanish. PMID 21757181
- [Background] Kueper T, Krohn M, Haustedt LO, Hatt H, Schmaus G, Vielhaber G. Inhibition of TRPV1 for the treatment of sensitive skin. Exp Dermatol. 2010 Nov;19(11):980-6. doi: 10.1111/j.1600-0625.2010.01122.x. PMID 20626462
- [Background] Stander S, Schneider SW, Weishaupt C, Luger TA, Misery L. Putative neuronal mechanisms of sensitive skin. Exp Dermatol. 2009 May;18(5):417-23. doi: 10.1111/j.1600-0625.2009.00861.x. PMID 19382311